CLINICAL TRIAL: NCT00530010
Title: A Humanitarian Device Exemption Use Protocol of TheraSphere for Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Radiolabeled Glass Beads in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NU 1365-001; P30CA060553 (NIH); NU-1365-001
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; advanced adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: yttrium Y 90 glass microspheres — The target dose of TheraSphere® is 80-150 Gy (8,000-15,000 rad). Patients may receive a single dose to the whole liver, or lobar treatment delivered as a sequence of treatments approximately 30 -90 days apart.

SUMMARY:
RATIONALE: Internal radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Using radiolabeled glass beads to kill tumor cells may be effective treatment for liver cancer that cannot be removed by surgery.

PURPOSE: This phase II trial is studying how well radiolabeled glass beads work in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide supervised access to treatment with yttrium Y 90 glass microspheres (TheraSphere®) to eligible patients with cancer of the liver who are not candidates for surgical resection.
* Evaluate patient experience and toxicities associated with yttrium Y 90 glass microspheres (TheraSphere®) treatment.

OUTLINE: This is a humanitarian device exemption use study.

Patients receive yttrium Y 90 glass microspheres (TheraSphere®) into the liver tumor through a percutaneously placed catheter into the hepatic artery. Patients may receive additional treatment 4-12 weeks after initial treatment at the discretion of the study physician.

After completion of study treatment, patients are followed at 2 weeks, 30 days, and then once a year for approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of intrahepatic carcinoma

  * Histopathology confirmation may be waived in patients with a radiographically identifiable liver mass AND known laboratory or clinical risk factors for cancer or elevated tumor markers such as AFP
* Unresectable disease
* No portal hypertension with portal venous shunt away from the liver
* No significant extrahepatic disease representing an imminent life-threatening outcome
* No evidence of potential delivery of > 16.5 mCi (30 Gy absorbed dose) radiation to the lungs on either of the following:

  * First yttrium Y 90 glass microspheres (TheraSphere®) administration
  * Cumulative delivery of radiation to the lungs over multiple treatments

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* Absolute granulocyte count ≥ 1,500/μL
* Platelet count > 25,000/μL
* Serum creatinine < 2.0 mg/dL (unless using non-iodinated contrast or on dialysis)
* Serum bilirubin ≤ 3.0 mg/dL (in some cases where there is an elevated bilirubin and the tumor may be isolated from a vascular standpoint, treatment may proceed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Any of the following contraindications to angiography and selective visceral catheterization:

  * History of severe allergy or intolerance to any contrast media, narcotics, sedatives, or atropine, that cannot be controlled using basic angiographic techniques
  * Bleeding diathesis, not correctable by usual forms of therapy
  * Severe peripheral vascular disease that would preclude catheterization
* Evidence of any detectable Tc-99 macroaggregated albumin flow to the stomach or duodenum, after application of established angiographic techniques to stop such flow
* Severe liver dysfunction or pulmonary insufficiency
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior and no other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable cancer primarily in the liver with the liver being the only site of disease or the dominant site of disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2004-12; Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Patient Completion | Through study completion, up to 24 months or when patient discontinues treatment for whatever reason.
  Proportion of patients completing scheduled treatment plan

CONTACTS AND LOCATIONS:
Overall Officials: Riad Salem, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Salem R, Lewandowski RJ, Mulcahy MF, Riaz A, Ryu RK, Ibrahim S, Atassi B, Baker T, Gates V, Miller FH, Sato KT, Wang E, Gupta R, Benson AB, Newman SB, Omary RA, Abecassis M, Kulik L. Radioembolization for hepatocellular carcinoma using Yttrium-90 microspheres: a comprehensive report of long-term outcomes. Gastroenterology. 2010 Jan;138(1):52-64. doi: 10.1053/j.gastro.2009.09.006. Epub 2009 Sep 18. PMID 19766639